CLINICAL TRIAL: NCT02316080
Title: Evaluating Remineralizers and Desensitizers Agents in Dental Bleaching Treatment: in Vitro and in Vivo Study
Brief Title: The Effect of Desensitizing Agents in In-home or In-office Dental Bleaching
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Camila Tirapelli, PhD, University of Sao Paulo
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Fapesp 2010120326
Record Dates: First submitted 2011-09-21; First posted 2014-12-12 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Dentin Hypersensitivity
Keywords: dental bleaching; dentin sensitivity; biomaterials
MeSH Terms: conditions — Dentin Sensitivity | interventions — tooth-bleaching agent, Opalescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Desensitizing therapy (Experimental): 14 groups (7 treated with in-office dental bleaching and 7 treated with home-use dental bleaching) . There will be 7 different types of dessensitizing agents that will be used together with the dental bleaching treatment
  Interventions: Other: Dental bleaching
- Dental Bleaching (Experimental): 2 groups of dental bleaching treatment - 16% carbamide peroxide and 35% peroxide
  Interventions: Other: Desensitizing therapy

INTERVENTIONS:
Other: Dental bleaching — Home-use or in-office dental bleaching was performed in patients that received different types od desensitizing therapy
  Other Names: Whitness Perfect®; Whitness HP®
  Arms: Desensitizing therapy
Other: Desensitizing therapy — Participants (in T1 and T2) used domestic-use (DU) or in office (IO) desensitizers (D): Control Group; (DU)- experimental dentifrice with 7,5% of Biosilicate micro-particles-(D1); Sensodyne® dentifrice-(D2); (DU)-Odontis RX Sensiblock® dentifrice-(D3); (IO)-Biosilicate micro-particles paste, 1:1-(D4); (IO)-bioglass type 45S5 paste, 1:1 (D6); (IO)-Desensebilize Nano P-(D6).
  Other Names: Dentifrice of Biosilicate; Sensodyne® dentifrice; Odontis RX Sensiblock; Biosilicate micro-particles paste, 1:1; Bioglass type 45S5 paste, 1:1; Desensebilize Nano P
  Arms: Dental Bleaching

SUMMARY:
The aim of this project is to evaluate in vitro and in vivo the effect of dental bleaching agents, carbamide peroxide 16% (T1) and hydrogen peroxide 35% (T2) together with desensitizers/remineralizer agents, Sensodyne® dentifrice (D1); experimental dentifrice with 7,5% of Biosilicate micro-particles (D2); Odontis RX® dentifrice (D3); Sorriso® dentifrice (D4); Biosilicate micro-particles paste, 1:1 (D5), Desensebilize Nano P (D6), bioglass type 45S5 paste, 1:1 (D7); GC= distilled water, in the experimental groups: T1/D1; T1/D2; T1/D3; T1/D4; T1/D5; T1/D6; T1/D7; T1/GC e T2/D1; T2/D2; T2/D3; T2/D4; T2/D5; T2/D6; T2/D7; T2/GC. In the in vitro study, microhardness and roughness measurements, and images using scanning electron microscopy (SEM) will be made on samples of bovine dental enamel and dentin (4x4x3mm; n=10 per group) before and after the treatment with the bleaching gels (T1= 14 days/ 04 hours/day; T2=single session) and the desensitizers/remineralizer agents. In the clinical study, the volunteers (n=10 per group) will be evaluated regarding dentin hypersensitivity (DH), using visual analogue scale, before the beginning of the treatments (T1 and T2) and during the next 14 days (1º, 3º, 7º, 10 º e 14º days) in which the desensitizers/remineralizer agents (there´s no control group in the clinical experiments) will be applying. Data will be analysed intra and inter-group, statistically.

DETAILED DESCRIPTION:
Background. Tooth sensitivity (TS) is a common side effect of tooth bleaching. The authors conducted a study to evaluate the efficiency of experimental desensitizing agents in reducing TS caused by bleaching agents.

Methods. To test experimental desensitizing agents in TS caused by dental bleaching the authors selected 113 participants without TS and randomly treated them with T1-16% carbamide peroxide (14 days) or T2-35% hydrogen peroxide (single session). The period of the study was 14 days. Participants (in T1 and T2) used domestic-use (DU) or in office (IO) desensitizers (D): Control Group; (DU)- experimental dentifrice with 7,5% of Biosilicate micro-particles-(D1); Sensodyne® dentifrice-(D2); (DU)-Odontis RX Sensiblock® dentifrice-(D3); (IO)-Biosilicate micro-particles paste, 1:1-(D4); (IO)-bioglass type 45S5 paste, 1:1 (D6); (IO)-Desensebilize Nano P-(D6). On days 1, 3, 7, 10 and 14, the authors received the participants to apply IO desensitizers and to record TS with Visual Analogue Scale (VAS). Data was analyzed with two-way ANOVA (considering time and desensitizing as factors) and post-hoc Bonferroni test (α=0.05).

Results. The use of experimental desensitizing agents G2 and G5 did not cause significantly difference in TS comparing to baseline. TS was not significantly different when G2 was used after 16% carbamide peroxide and G5 after 35% hydrogen peroxide application. Self-perception TS values were significantly (p<0.001) higher than recorded VAS.

Conclusions. Experimental desensitizing agents containing Biosilicate® can prevent TS caused by bleaching agents: in dentifrice form when associated to 16% carbamide peroxide and in paste, when 35% hydrogen peroxide is used.

ELIGIBILITY:
Inclusion Criteria:

1. Patients male or females, aged between 18 and 40 years.
2. Smokers and nonsmokers.
3. Patients with good general health.
4. Patients with good oral health (no changes in hard or soft tissues).
5. Have a minimum of 24 permanent teeth present and no restorations on anterior teeth.

Exclusion Criteria:

1. Patients with a medical history marked by chronic use of analgesics, anti-inflammatory and psychotropic drugs.
2. Patients with braces or prostheses or restorations on anterior teeth.
3. Patients with periodontal disease or poor oral hygiene.
4. Patients with prior tooth sensitivity or have made use of desensitizing agents in the last three months.
5. Patients who are pregnant or nursing.
6. Patients with eating disorders or dieting too acidic.
7. Systemic conditions that predispose to tooth sensitivity.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Dentin hypersensitivity | Baseline
  The pain caused by dentin hypersensitivity was measured by stimulating cervical region of the teeth with a blast of air from a triple seringe and the patient will relate his/her pain in accordance with a visual analog scale (VAS) which consists of a 1 to 10 scale where the patients recorded their dentin hypersensitivity when stimulated. Dentin hypersensitivity (DH) was measured, using visual analogue scale, before the beginning of the treatments (baseline -T1 and T2) and during the next 14 days (1º, 3º, 7º, 10 º e 14º days)

SECONDARY OUTCOMES:
Dentin hypersensitivity | Day 1
  The pain caused by dentin hypersensitivity was measured by stimulating cervical region of the teeth with a blast of air from a triple seringe and the patient will relate his/her pain in accordance with a visual analog scale (VAS) which consists of a 1 to 10 scale where the patients recorded their dentin hypersensitivity when stimulated. Dentin hypersensitivity (DH) was measured, using visual analogue scale, before the beginning of the treatments (baseline -T1 and T2) and during the next 14 days (1º, 3º, 7º, 10 º e 14º days)
Dentin hypersensitivity | Day 3
  The pain caused by dentin hypersensitivity was measured by stimulating cervical region of the teeth with a blast of air from a triple seringe and the patient will relate his/her pain in accordance with a visual analog scale (VAS) which consists of a 1 to 10 scale where the patients recorded their dentin hypersensitivity when stimulated. Dentin hypersensitivity (DH) was measured, using visual analogue scale, before the beginning of the treatments (baseline -T1 and T2) and during the next 14 days (1º, 3º, 7º, 10 º e 14º days)
Dentin hypersensitivity | Day 7
  The pain caused by dentin hypersensitivity was measured by stimulating cervical region of the teeth with a blast of air from a triple seringe and the patient will relate his/her pain in accordance with a visual analog scale (VAS) which consists of a 1 to 10 scale where the patients recorded their dentin hypersensitivity when stimulated. Dentin hypersensitivity (DH) was measured, using visual analogue scale, before the beginning of the treatments (baseline -T1 and T2) and during the next 14 days (1º, 3º, 7º, 10 º e 14º days)
Dentin hypersensitivity | Day 10
  The pain caused by dentin hypersensitivity was measured by stimulating cervical region of the teeth with a blast of air from a triple seringe and the patient will relate his/her pain in accordance with a visual analog scale (VAS) which consists of a 1 to 10 scale where the patients recorded their dentin hypersensitivity when stimulated. Dentin hypersensitivity (DH) was measured, using visual analogue scale, before the beginning of the treatments (baseline -T1 and T2) and during the next 14 days (1º, 3º, 7º, 10 º e 14º days)
Dentin hypersensitivity | Day 14
  The pain caused by dentin hypersensitivity was measured by stimulating cervical region of the teeth with a blast of air from a triple seringe and the patient will relate his/her pain in accordance with a visual analog scale (VAS) which consists of a 1 to 10 scale where the patients recorded their dentin hypersensitivity when stimulated. Dentin hypersensitivity (DH) was measured, using visual analogue scale, before the beginning of the treatments (baseline -T1 and T2) and during the next 14 days (1º, 3º, 7º, 10 º e 14º days)

CONTACTS AND LOCATIONS:
Overall Officials: Camila Tirapelli, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo -Ribeirao Preto Campus, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- See also: Dental School of Ribeirao Preto website — http://www.forp.usp.br/